CLINICAL TRIAL: NCT04836806
Title: Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy of Cetirizine and Famotidine in Reducing the Duration of Symptoms in Patients With COVID-19: A Pilot Study
Brief Title: Cetirizine and Famotidine for COVID-19
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to issues with enrollment and lack of funding.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Humphrey Lam, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001722
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Cetirizine; Famotidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cetirizine and famotidine (Experimental): Participants testing positive for COVID-19 who are randomized to take cetirizine and famotidine for 10 days.
  Interventions: Drug: Cetirizine and Famotidine
- Placebo (Placebo Comparator): Participants testing positive for COVID-19 who are randomized to take a placebo to match cetirizine and famotidine for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cetirizine and Famotidine — Participants will take 10 milligrams (mg) of cetirizine once a day and 20 mg of famotidine twice a day for 10 days (two pills in the morning and one in the evening).
  Other Names: Zyrtec; Pepcid
  Arms: cetirizine and famotidine
Drug: Placebo — Participants will take placebos to match 10 mg of cetirizine once a day and 20 mg of famotidine twice a day for 10 days (two pills in the morning and one in the evening).
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial to evaluate the efficacy of cetirizine and famotidine in reducing the duration of symptoms in patients with COVID-19. Secondary aims are to determine if cetirizine and famotidine decrease severity and duration of symptoms, incidence of hospitalizations, ICU admissions, and death.

DETAILED DESCRIPTION:
COVID-19 is a disease caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Patients with COVID-19 may present with a myriad of symptoms ranging from fever and cough to more severe symptoms such as shortness of breath. Cetirizine and famotidine are commonly administered medications that can be found over-the-counter. They are well tolerated and have low potential for drug-drug interaction. With it's anti-inflammatory properties via modulation of proinflammatory cytokines, cetirizine may be an effective symptomatic therapeutic for COVID-19. With possible antiviral properties, famotidine may have a role in therapy as well.

After a positive COVID test has been confirmed, participants with be randomized to take cetirizine and famotidine or a placebo for 10 days and the study medication will be shipped to them. Participants will record their symptoms for 30 days and any serious adverse events will be followed for up to 60 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* positive COVID-19 test (antigen or PCR)
* symptomatic from COVID-19
* symptoms less than or equal to 7 days

Exclusion Criteria:

* already enrolled in another COVID-19 drug study
* chronically taking a H1-receptor antagonist or H2-receptor antagonist
* have taken H1-receptor antagonist or H2-receptor antagonist less than 72 hours from expressed interest in the study.
* history of an adverse reaction to H1 or H2-receptor antagonists
* severe liver disease
* severe renal disease
* taking steroids
* taking hydroxychloroquine and/or azithromycin
* already participating in a COVID-19 vaccine trial
* already received a COVID-19 vaccine
* symptoms greater than 7 days
* have had COVID-19 more than once

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of symptoms | Day 30
  Participants will record their oral temperature and the presence of COVID-19 symptoms of cough, shortness of breath/difficulty breathing, fatigue, myalgias, headache, loss of taste, loss of smell, sore throat, rhinorrhea, congestion, nausea/vomiting, diarrhea, and feverishness/chills, twice daily for up to 14 days. The number of days until resolution of overall symptoms of COVID-19 will be compared between study arms.

SECONDARY OUTCOMES:
Severity of Symptoms | Day 30
  Participants will record their severity of COVID-19 symptoms of cough, shortness of breath/difficulty breathing, fatigue, myalgias, headache, loss of taste, loss of smell, sore throat, rhinorrhea, congestion, nausea/vomiting, diarrhea, and feverishness/chills on a four-point scale (where 0 = absent, 1 = mild, 2 = moderate, and 3 = severe) twice daily for up to 14 days.
Time to Resolution of Individual Symptoms | Day 30
  Participants will record their oral temperature and the presence of COVID-19 symptoms of cough, shortness of breath/difficulty breathing, fatigue, myalgias, headache, loss of taste, loss of smell, sore throat, rhinorrhea, congestion, nausea/vomiting, diarrhea, and feverishness/chills, twice daily for up to 14 days. The number of days until resolution of individual symptoms of COVID-19 will be compared between study arms.
Incidence of Hospitalization | Day 30
  Hospitalizations will be compared between study arms.
Incidence of Intensive Care Unit (ICU) Admission | Day 60
  Admissions to the ICU will be compared between study arms.
Incidence of Death | Day 60
  The number of deaths will be compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Humphrey Lam, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital at Wesley Woods COVID-19 Testing Facility, Atlanta, Georgia
  - Emory Healthcare Network Peachtree Immediate Care COVID-19 Testing Centers, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No